CLINICAL TRIAL: NCT06472141
Title: Effectiveness of Cervical Stabilization Exercises in Individuals With Temporomandibular Joint Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Mesut Arslan, Assistant Professor, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMJD-EXERCISE
Record Dates: First submitted 2024-06-10; First posted 2024-06-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This study was planned as a randomized controlled trial. The individuals included in the study will be divided into 2 groups as Stabilization and Control group by block randomization method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group will receive a standard treatment (education + home exercises) program.
  Interventions: Other: Standard treatment (Education + home exercises)
- Stabilization group (Experimental): The stabilization group will receive cervical stabilization exercises in addition to standard treatment.
  Interventions: Other: Cervical stabilization exercises; Other: Standard treatment (Education + home exercises)

INTERVENTIONS:
Other: Cervical stabilization exercises — Cervical Stabilization Exercises will be performed 3 days a week for 8 weeks.
  Arms: Stabilization group
Other: Standard treatment (Education + home exercises) — Individuals will be informed about TMJ disorders, parafunctional activities (chewing gum, nail/pen biting, etc.) and recommendations. In addition, Rocabado exercises will be given as a home program.

SUMMARY:
It is planned to examine the effect of cervical stabilization exercises on Temporomandibular Joint (TMJ) symptoms in individuals with TMJ disorder.

DETAILED DESCRIPTION:
Individuals included in the study will be divided into 2 groups, Stabilization and Control groups, by block randomization method. A standard treatment program (Education + home exercises) will be applied to both groups. In addition to the stabilization group, cervical stabilization exercises will be applied. Individuals will be evaluated with the Sociodemographic Data Form before the application.

Before and after the application, individuals were assessed for TMJ pain with the Numeric Pain Rating Scale (NPRS), TMJ symptom severity with the Fonseca Anamnestic Index (FAI) and cervical posture, mobility and muscle performance will be evaluated with craniovertebral angle, goniometer and craniocervical flexion test.

ELIGIBILITY:
Inclusion Criteria:

* Having a TMJ disorder according to the TMJ Disorders Research Diagnostic Criteria (RDC/TMD),
* Being between the ages of 18-65,

Exclusion Criteria:

* Neurological diseases (such as Multiple Sclerosis, Parkinson's disease),
* Metabolic and systemic diseases (such as Hypothyroidism, Hypercalcemia, Diabetes mellitus, Celiac disease),
* Rheumatologic diseases (such as Rheumatoid arthritis, Scleroderma),
* History of head and spine trauma/surgery in the last 6 months,
* History of malignancy and pregnant women will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Change from baseline at 8 weeks
  TMJ pain will be evaluated at rest with the NPRS scale. It is a scale scored between 0-10 points and '0 points means 'I have no pain' and '10 points means 'I have unbearable pain'. NRS score between 1-3 points indicates mild pain, between 4-6 points indicates moderate pain and between 7-10 points indicates severe pain.
Fonseca Anamnestic Index (FAI) | Change from baseline at 8 weeks
  It assesses TMJ disorder and its severity. The index includes three options: "yes" (10 points), "sometimes" (5 points) and "no" (0 points). A total score of 0-15 is considered as no TMJ disorder, 20-40 as mild, 45-65 as moderate, and 70-100 as severe.
Cervical Posture | Change from baseline at 8 weeks
  Cervical posture will be evaluated from the craniovertebral angle.
Cervical Mobility | Change from baseline at 8 weeks
  For cervical mobility, normal joint movements of the neck will be evaluated with a goniometer.
Cervical Muscle Performance | Change from baseline at 8 weeks
  Cervical muscle performance will be evaluated with the craniocervical flexion test.

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis Eren Üniversitesi, Merkez, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No